CLINICAL TRIAL: NCT05361083
Title: Studies of 18F-CETO as a Tracer for Adrenal PET Diagnostics
Brief Title: First-in-human Evaluation of [18F]CETO
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other); British Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-004831-64
Record Dates: First submitted 2022-04-22; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Primary Aldosteronism Due to Aldosterone Producing Adenoma; Primary Aldosteronism Due to Nodular Hyperplasia; Adrenal Cushing Syndrome; Non-Secretory Adrenal Adenoma; Adrenocortical Carcinoma
MeSH Terms: conditions — ACTH Syndrome, Ectopic; Adrenocortical Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- First-in-man investigastion of [18F]CETO (Experimental): 15 patients were investigated with PET/CT after injection of 2,5 MBq/kg [18F]CETO. 5 healthy volunteers were investigated twice (Test-retest), with approximately 2 weeks in-between each PET/CT investigation, after injection of 1,3 MBq/kg [18F]CETO. Arterial blood samples were taken as well as urinary sampels.
  3 out of 5 healthy volunteers were also investigated twice with PET/CT after injection of 13,2 MBq/kg [15O]water, performed before the [18F]CETO PET/CT.
  Interventions: Drug: F18CETO

INTERVENTIONS:
Drug: F18CETO — Injection of F18CETO or O15water followed by PET/CT
  Other Names: Para-chloro-2-[18F]fluoroethyletomidate

SUMMARY:
Purpose of this clinical phase 1 trial was to determine if para-chloro-2-[18F]fluoroethyletomidate positron emission computed tomography ([18F]CETO-positron emission computed tomography(PET)/computed tomography(CT)) can be used in diagnostics of adrenal tumors and if the biochemical/pharmacological states conditions in humans with various illnesses, compared to healthy humans, such as the radio tracer is suitable?

DETAILED DESCRIPTION:
After receiving oral and written information about the study and its potential risks, all participants provided written informed consent. All participants underwent a screening visit 1-28 days before their [18F]CETO PET/CT. At the screening visit their medical history was obtained, including besides information of previous disease(s) and medication, also a clinical examination, WHO performance status, height, weight, pulse rate and blood pressure, blood chemistry and haematology.

Right before the PET/CT investigation a baseline assessment was performed including:

* A physical examination according to Modified Early Warning Score (MEWS)
* 12-lead electrocardiogram (ECG)
* Any concomitant medications was recorded
* Medical history - occurrence of any new symptoms and events since the screening visit
* Hematology (International Normalized Ratio (INR) in patients with antiocoagulant treatment).
* Pregnancy test in women.
* Assessment of injection site monitored by visual inspection (rash and phlebitis)

Participants received on average 0,76 mikrograms (range 0,1-1.37 mikrograms) of administered mass of CETO in conjunction to the PET/CT investigation.

Potential adverse events were monitored closely during, and after the administration of [18F]CETO, with access to emergency medicine resources.

Each participant remained for observation at least 3 hours after administration of [18F]CETO and the following assessments were performed:

* Blood withdrawn for additional post-scan chemical analysis.
* Assessment of injection site monitored by visual inspection (rash and phlebitis).
* MEWS

The ten first participants were evaluated for serious adverse events/adverse events (SAE/AEs) the day after (approximately 24 hours after) performing the [18F]CETO PET due to the short half-life of the radionuclide used, fluorine- 18 (T1/2= 109.5 min). Safety reporting was assessed by use of clinical Adverse Events and Common Toxicity Criteria (CTC), laboratory and non-laboratory toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with adrenal incidentalomas with an concurrent overproduction of aldosterone or cortisol or no concurrent hormone production, or patients diagnosed with adrenocortical carcinoma
* For healthy volunteers inclusion criteria included no known diseases, no ongoing medication and no known adrenal anomalies.

Exclusion Criteria for patients and healthy volunteers:

* pregnancy, age below 18, claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Evaluate safety of up to two administrations of [18F]CETO in up to 15 patients in comparison with 5 healthy controls. | Up to 1 day after the [18F]CETO PET/CT for each patient
  Number of patients with treatment-related adverse events as assessed by clinical Adverse Events and Common ToxicityNCI Common Terminology Criteria for Adverse Events v4.0 (CTCAE)

SECONDARY OUTCOMES:
Evaluate [18F]CETO as a PET- biomarker for the adrenals and to diagnose and visualize primary aldosteronism, cortisol producing adrenocortical adenoma and non-functioning adrenocortical adenoma in up to 15 patients | Up to 24 month
  Arterial blood was collected to determined the fraction of intact [18F]CETO in plasma. PET- modelling based on dynamic PET-data and metabolite analysis was performed for scientific purposes. Measurement of Standard Uptake Value (SUV) was determined for the adrenal glands.
Biodistribution of [18F]CETO | Up to 22 month
  Measurement of SUV for organs was determined.
Compare uptake of [18F]CETO in normal adrenal glands in patients comparing healthy controls and determine the test - retest variability of [18F]CETO. | Up to 24 month
  Difference in SUV in the adrenal glands between two investigations in the samt participant was determined.

CONTACTS AND LOCATIONS:
Overall Officials: Per Hellman, Professor, Study Director — Uppsala University and Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silins I, Moreno A, Wall A, Aigbirhio F, Gurnell M, Brown M, Roslin S, Antoni G, Hellman P, Sundin A, Lubberink M. Radiation dosimetry of para-chloro-2-[18F]fluoroethyl-etomidate: a PET tracer for adrenocortical imaging. EJNMMI Res. 2024 May 21;14(1):48. doi: 10.1186/s13550-024-01109-2. PMID 38771379
- [Derived] Silins I, Sundin A, Lubberink M, O'Sullivan L, Gurnell M, Aigbirhio F, Brown M, Wall A, Akerstrom T, Roslin S, Hellman P, Antoni G. First-in-human evaluation of [18F]CETO: a novel tracer for adrenocortical tumours. Eur J Nucl Med Mol Imaging. 2023 Jan;50(2):398-409. doi: 10.1007/s00259-022-05957-9. Epub 2022 Sep 8. PMID 36074157